CLINICAL TRIAL: NCT05080452
Title: Visualizing Anterior Cutaneous Nerve Entrapment Syndrome (ACNES) and Lumbar Cutaneous Nerve Entrapment Syndrome (LUCNES) With Dynamic Infrared Thermography (DIRT)
Brief Title: Visualizing ACNES and LUCNES With DIRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: Coming
Record Dates: First submitted 2019-07-26; First posted 2021-10-15 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Nerve Compression Syndrome; Abdominal Pain; Lower Back Pain
Keywords: Thermography; CT angiography; Color Doppler
MeSH Terms: conditions — Nerve Compression Syndromes; Abdominal Pain; Low Back Pain | interventions — Computed Tomography Angiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACNES patients: Patients referred to ultrasound-guided treatment for abdominal wall pain caused by ACNES
  Interventions: Diagnostic Test: Dynamic infrared thermography (DIRT)
- LUCNES patients: Patients referred to ultrasound-guided treatment for lower back pain caused by LUCNES
  Interventions: Diagnostic Test: Dynamic infrared thermography (DIRT)

INTERVENTIONS:
Diagnostic Test: Dynamic infrared thermography (DIRT) — Visualizing hot spots
  Other Names: Comparison to color Doppler ultrasound and CT angiography

SUMMARY:
Anterior cutaneous nerve entrapment syndrome (ACNES) is caused by nerve entrapment in the abdominal wall. Recently de Weerd and Weum have suggested lumbar cutaneous nerve entrapment syndrome (LUCNES) as a name for a similar condition in the lower back. DIRT can potentially be used to identify the locations of perforators, thereby also indirectly identifying the location of nerve entrapment in ACNES and LUCNES, when a point of maximal pain corresponds to a hot spot. This study evaluates the location of hot spots on DIRT in relation to tender points and perforators visualized with CT angiography and color Doppler. In the ACNES patients, DIRT performed with a low-cost smartphone thermal camera will be compared to DIRT with a professional thermal camera to evaluate the usefulness of low-cost equipment to visualize the point of nerve entrapment.

DETAILED DESCRIPTION:
Background

Anterior cutaneous nerve entrapment syndrome (ACNES) is caused by nerve entrapment in the abdominal wall. The entrapment is believed to occur at the exit point of the sensate nerve through the anterior fascia of the rectus abdominis muscle. The diagnosis is mainly based on patient history and clinical examination. Pain relief after local anaesthesia may support the diagnosis. Often patients go through many diagnostic procedures to exclude other possible causes of abdominal pain. In such, ACNES is often an exclusion diagnosis. Recently Weum and de Weerd published an article describing perforator-guided treatment of ACNES using botulinum toxin serotype A (BTA). Based on anatomical knowledge and clinical experience, they used color Doppler ultrasound (CDU) to visualize the vascular structures called perforators that accompany the nerves at the exit points through the anterior rectus fascia. They noticed that accurate placement of the needle at this exit point triggered the same pain as caused by ACNES. Their earlier publications on dynamic infrared thermography (DIRT) in perforator mapping show that the locations of perforators can be visualised as hot spots on the abdominal skin.

Based on their experimental and clinical experience, they found that lower back pain might be caused by nerve entrapment, similar as seen in ACNES. In a pilot study using CDU, they found that the point of maximal pain, as marked by the patient, corresponded with the exit point of a perforator through the lumbar fascia. Knowledge from the use of a lumbar artery perforator flap makes it very likely that the sensate nerve accompanies these perforator vessels. Recently de Weerd and Weum have suggested lumbar cutaneous nerve entrapment syndrome (LUCNES) as a name for this condition. DIRT can potentially be used to identify the locations of these perforators, thereby also indirectly identifying the location of nerve entrapment, when a point of maximal pain corresponds to a hot spot.

Although DIRT has been used in several patients as an adjunct to support the diagnosis of ACNES, there are no studies that have systematically evaluated the use of DIRT in the diagnosis of ACNES or LUCNES. If DIRT could contribute to confirm the diagnosis ACNES or LUCNES, such would be valuable for clinicians as well as patients. Today, ACNES is often a diagnosis made by excluding other causes of pain. If DIRT can be used a reliable technique in the diagnosis of ACNES and LUCNES, such would be of great psychological value to the patients and may contribute to reduced health care costs.

General practitioners are often the first health care providers that see patients with abdominal wall pain and lower back pain. Reliable perforator mapping with DIRT has until recently only been possible with expensive professional thermography equipment. Low-cost thermography cameras for smartphones are now available. If these cameras can provide reliable information on the location of perforators, and thereby also the location of nerve entrapment, general practitioners and other clinicians could use DIRT as a diagnostic tool for this patient group without expensive professional thermography equipment.

Aim and hypotheses

The aim of the study is to evaluate the usefulness of DIRT in the diagnostics of ACNES and LUCNES, as well as evaluating if inexpensive smartphone thermal cameras are equally reliable as professional thermography equipment in the diagnostics of ACNES.

Hypothesis 1: DIRT is a reliable tool to support the diagnosis of ACNES.

Hypothesis 2: DIRT is a reliable tool to support the diagnosis of LUCNES.

Hypothesis 3: Smartphone thermal cameras are equally reliable as professional thermography equipment in the diagnosis of ACNES.

Materials and methods

Patients will be recruited on a voluntary basis from the list of patients referred to the outpatient clinic at the department of plastic surgery, University hospital of North Norway (UNN), with the diagnosis ACNES or LUCNES. Only patients above the age of 18 years, that are not pregnant, with no history of allergic reactions to iodine contrast media, reduced renal function or kidney disease will be included. Based on clinical experience and previous research on perforator mapping, we estimate that 25 patients from each group will provide reliable data to evaluate the usefulness of DIRT.

Patients will be instructed to mark the location of maximal pain on their abdominal wall (ACNES) or lower back (LUCNES) with a permanent marker before arrival at the outpatient clinic. DIRT will be performed simultaneously with professional thermography equipment and a smartphone thermal camera, using the protocol described by Weum and de Weerd. Afterward the point of maximal pain will be marked with a plastic marker taped to the skin, before CTA is performed in the arterial phase. ACNES patients are examined in the supine position, and LUCNES patients in the prone position. The student will perform CDU to evaluate if the point of maximal pain corresponds with a perforator exiting the muscle fascia.

All patients recruited are referred to ultrasound-guided injection with BTA. If CDU reveals that the point of maximal pain corresponds to the exit point of a perforator, the student will perform an ultrasound-guided injection of BTA around the perforator at the exit point. The student will collect data about pain related to needle placement and injection of BTA.

All data will be analyzed with respect to the reliability of DIRT, both with professional equipment and smartphone thermal camera, to identify the location of nerve entrapment. As DIRT only provides indirect information on the point of nerve entrapment, the findings from DIRT will be compared with the findings from both CTA and CDU, which are imaging modalities that are able to visualize these exit points accurately. As an indicator of the usefulness of DIRT, the student will also evaluate the effect of BTA on the pain reported by patients three weeks after the procedure using a VAS score and quality of life assessment compared with data collected before the treatment.

As all patients have been referred for ambulatory treatment at UNN, clinical data will be stored in the electronic patient journal. Findings from the imaging modalities will be stored in the RIS and PACS system at the department of radiology. Following approval by the data protection officer at UNN, depersonalized data will be stored at secure research server and used for later analysis. Data will be stored for seven years after publication and then deleted.

ELIGIBILITY:
Inclusion Criteria:

ACNES and LUCNES patients referred for ambulatory ultrasound-guided treatment

Exclusion Criteria:

Former reaction to contrast media used for CT angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 patients with clinical signs of ACNES 25 patients with clinical signs of LUCNES
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison tender spot coordinates and DIRT coordinates with professional thermocamera | One day
  Distance between coordinates (cm) to evaluate agreement
Comparison tender spot coordinates and CT angiography coordinates | One day
  Distance between coordinates (cm) to evaluate agreement
Comparison tender spot coordinates and color Doppler coordinates | One day
  Distance between coordinates (cm) to evaluate agreement
Comparison hot spot coordinates smarphone/professional thermocamera | One day
  Evaulation if same hot spots are visible on thermal images from both cameras

CONTACTS AND LOCATIONS:
Overall Officials: Sven Weum, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindsetmo RO, Stulberg J. Chronic abdominal wall pain--a diagnostic challenge for the surgeon. Am J Surg. 2009 Jul;198(1):129-34. doi: 10.1016/j.amjsurg.2008.10.027. PMID 19555786
- [Background] Weum S, de Weerd L. Perforator-Guided Drug Injection in the Treatment of Abdominal Wall Pain. Pain Med. 2016 Jul;17(7):1229-32. doi: 10.1093/pm/pnv011. Epub 2015 Dec 7. PMID 26814247
- [Background] Weum S, Mercer JB, de Weerd L. Evaluation of dynamic infrared thermography as an alternative to CT angiography for perforator mapping in breast reconstruction: a clinical study. BMC Med Imaging. 2016 Jul 15;16(1):43. doi: 10.1186/s12880-016-0144-x. PMID 27421763
- [Background] de Weerd L, Weum S, Mercer JB. The value of dynamic infrared thermography (DIRT) in perforatorselection and planning of free DIEP flaps. Ann Plast Surg. 2009 Sep;63(3):274-9. doi: 10.1097/SAP.0b013e3181b597d8. PMID 19700958
- [Background] de Weerd L, Weum S. The butterfly design: coverage of a large sacral defect with two pedicled lumbar artery perforator flaps. Br J Plast Surg. 2002 Apr;55(3):251-3. doi: 10.1054/bjps.2002.3791. PMID 12041981
- [Background] de Weerd L, Elvenes OP, Strandenes E, Weum S. Autologous breast reconstruction with a free lumbar artery perforator flap. Br J Plast Surg. 2003 Mar;56(2):180-3. doi: 10.1016/s0007-1226(03)00039-0. PMID 12791371
- [Background] Weum S, Lott A, de Weerd L. Detection of Perforators Using Smartphone Thermal Imaging. Plast Reconstr Surg. 2016 Nov;138(5):938e-940e. doi: 10.1097/PRS.0000000000002718. No abstract available. PMID 27783018
- [Background] Cina A, Salgarello M, Barone-Adesi L, Rinaldi P, Bonomo L. Planning breast reconstruction with deep inferior epigastric artery perforating vessels: multidetector CT angiography versus color Doppler US. Radiology. 2010 Jun;255(3):979-87. doi: 10.1148/radiol.10091166. Epub 2010 Apr 14. PMID 20392982